CLINICAL TRIAL: NCT06333041
Title: Randomized, Double-Blind, Placebo-Controlled Cross-Over Study to Evaluate the Effects of Cannabidiol on Neurobehavioral and Function Outcomes in Sanfilippo Syndrome
Brief Title: Study of Cannabidiol in Sanfilippo Syndrome
Status: Not yet recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center (Other)
Responsible Party: Principal Investigator, Lynda E Polgreen, Associate Professor of Pediatrics, Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 32977-01-00
Record Dates: First submitted 2024-03-20; First posted 2024-03-27 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2024-10

CONDITIONS: Sanfilippo Syndrome; Mucopolysaccharidosis III
Keywords: Cannabidiol; Epidiolex
MeSH Terms: conditions — Mucopolysaccharidosis III | interventions — Cannabidiol

STUDY DESIGN:
Intervention Model Description: Double-blind, placebo-controlled, cross-over study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Epidiolex (cannabidiol) (Experimental): Oral Epidiolex (cannabidiol) administered twice daily (BID) Week 1: 5 mg/kg/day BID Weeks 2-8: 10 mg/kg/day BID Weeks 9-16: 20 mg/kg/day BID
  8-week washout; cross-over to placebo comparator starting on Week 24.
  Interventions: Drug: Epidiolex
- Placebo (PBO) (Placebo Comparator): Week 1: Dose escalate to maximum tolerated placebo dose Weeks 2-16: Maximum tolerated placebo dose
  8-week washout; cross-over to Experimental group starting at week 24, following the same dose-escalation as the Experimental arm.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Epidiolex — Epidiolex (cannabidiol) oral solution is a clear, colorless to yellow liquid containing cannabidiol at a concentration of 100 mg/mL. Inactive ingredients include dehydrated alcohol (7.9% w/v), sesame seed oil, strawberry flavor, and sucralose.
  Other Names: Cannabidiol; CBD
  Arms: Epidiolex (cannabidiol)
Drug: Placebo — Placebo oral solution is a yellow oily solution containing the excipients sesame oil and anhydrous ethanol with added sweetener (sucralose) and strawberry flavoring
  Arms: Placebo (PBO)

SUMMARY:
The goal of this clinical trial is to test cannabidiol in Sanfilippo syndrome. The main questions it aims to answer are: 1) determine the safety of cannabidiol in Sanfilippo syndrome, and 2) explore the efficacy of cannabidiol in treating the neurobehavioral symptoms and functional outcomes of Sanfilippo syndrome.

Each participant's caregiver will be asked to complete surveys related to the participant's behavior, mood, sleep, stooling, pain, and caregiver stress intermittently throughout the study. All participants will be enrolled into one of two cohorts based on enrollment order:

1. Sentinel Safety Cohort (first 5 participants) - all participants treated with Epidiolex (cannabidiol)
2. Controlled Cohort (next 30 participants) - participants randomized 1:1 (equal chance) to start treatment with Epidiolex (cannabidiol) or placebo for 16 weeks, followed by an 8-week washout period (no treatment). Participants then switch to the opposite treatment group for 16 weeks followed by all participants treated for 52 weeks with Epidiolex (cannabidiol).

DETAILED DESCRIPTION:
Sanfilippo syndrome, or Mucopolysaccharidosis type III (MPS III), is a rare genetic lysosomal storage disease characterized by the accumulation of heparan sulfate due to insufficient production of lysosomal enzymes. Consequently, a buildup of heparan sulfate causes progressive neurodegeneration, leading to significant neurobehavioral problems. These neurobehavioral symptoms are highly disruptive and distressing to families, have a significant impact on the quality of life of the patients and their families, and likely interfere with adjunctive therapeutic attempts at supporting the child. To date, there are no approved therapies for the treatment of the neurobehavioral symptoms of Sanfilippo syndrome. Cannabidiol (CBD), a compound derived from the cannabis plant but without the psychoactive effects, has been shown to be safe and effective in the treatment of children with severe epilepsy disorders. Studies have shown that CBD improves behavior in children with autism. This study will use Epidiolex, a pharmaceutical-grade purified oral solution of cannabidiol that was approved by the FDA for the treatment of severe pediatric epilepsy disorders. Study subjects will include approximately 35 participants with Sanfilippo syndrome. Participants will undergo baseline clinical evaluations, and neurobehavioral, and functional outcomes will be collected from parent-reported questionnaires. Participants will then receive either Epidiolex or placebo for 16 weeks. Following this period and an 8-week washout, participants will cross over and receive the opposite treatment for 16 weeks. Safety labs and questionnaires will be collected throughout these periods to assess safety and efficacy. Participants and study personnel will be blinded to the treatment status of each participant. When this blinded portion of the trial is completed, all participants will receive Epidiolex open-label for 52 weeks to measure long-term safety. The type and severity of adverse events will be collected to measure safety, and different behavioral and functional outcomes will be collected to measure efficacy.

ELIGIBILITY:
Inclusion Criteria:

* MPS III diagnosis confirmed by genetic testing
* ≥ 4 years of age
* Patient or parent/legal guardian is able and willing to provide informed consent. For patients 7 to 16 years of age, assent must also be provided when cognitively possible.
* If taking any of the following, no dose changes for the last 8 weeks:

  1. Anakinra
  2. Fluoxetine
  3. Probiotic supplement
* One of the following criteria are met:

  1. Previous participation in a gene/cell therapy or enzyme restorative clinical trial.
  2. Previously ineligible to participate in a gene/cell therapy or enzyme restorative clinical trial due to advanced disease state.
  3. Functional age, as measured by the Vineland, is ≤ 0.5 chronological age

Exclusion Criteria:

Equitable selection will be used when choosing participants. An individual who meets any of the following criteria will be excluded from participation in this study:

* Mutation known to cause slowly progressive disease
* Taken any form of cannabis, including cannabidiol, in the last 8 weeks
* Currently enrolled in another ongoing clinical trial
* Concomitant use of any of the following therapies:

  * Rifampin
  * Diazepam (except for intermittent use as needed for treatment of a prolonged seizure episode)
  * Clobazam
  * Stiripentol
  * Everolimus, sirolimus, tacrolimus
  * Digoxin
  * Valproate
  * Recreational or medical Tetrahydrocannabinol (THC) or synthetic cannabinoid medications (including Sativex) within the last three months
  * Felbamate (if taking for less than one year)
* Non-pharmacological therapies (e.g. ketogenic diet) must be stable for up to four weeks prior to enrollment
* Clinical evidence of liver disease or liver injury as indicated by the presence of abnormal tests (AST or ALT > 2 x ULN; Bilirubin > 2 x ULN)
* Known hypersensitivity to any components of Epidiolex (cannabidiol)
* Pregnant or lactating women
* Any other social or medical condition that the investigator believes would pose a significant hazard to the subject if the investigational therapy were initiated or be detrimental to the study

Min Age: 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2025-06 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Sanfilippo Behavior Rating Scale (SBRS)- mood/anger/aggression score | Changes over 16 weeks of treatment versus 16 weeks of placebo
  The Sanfilippo Behavior Rating Scale is a 68-item questionnaire, developed by Shapiro et al to assess the behavioral phenotype of children with Sanfilippo syndrome and its progression over time. The Sanfilippo Behavior Rating Scale mood/anger/aggression cluster is one of four clusters and two domains that make up the Sanfilippo Behavior Rating Scale. A higher score indicates more severe mood/anger/aggression symptoms. Each question within the mood/anger/aggression cluster is scored on a scale of 0-6 and a total mean score is calculated. The mean mood/anger/aggression score is standardized using the mean and standard deviation from a cohort of Sanfilippo patients, categorized as "slow progressors," ages 81-220 months. This reference cohort was chosen to best match the age distribution of our participants.

CONTACTS AND LOCATIONS:
Locations (1):
- The Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center, Torrance, California, United States

IPD SHARING:
Plan to Share IPD: No